CLINICAL TRIAL: NCT01460771
Title: Pilot Open-label and Blinded Clinical Trial of Transcranial Direct-current Stimulation in Childhood Dystonia
Brief Title: Transcranial Direct-Current Stimulation in Childhood Dystonia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Crowley Carter Foundation (Other); Don and Linda Carter Foundation (Other)
Responsible Party: Principal Investigator, Terence Sanger, Associate Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDCS2011
Record Dates: First submitted 2011-09-27; First posted 2011-10-27 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Childhood Onset Dystonias
Keywords: childhood dystonia
MeSH Terms: conditions — Dystonic Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Active Transcranial Direct Current Stimulation (TDCS) at 1mA or highest tolerated current
  Interventions: Device: TDCS (Transcranial Direct-current Stimulation)
- sham (Sham Comparator): inactive Transcranial Direct current stimulation (TDCS) at 0mA
  Interventions: Device: sham TDCS (Transcranial Direct-current Stimulation)

INTERVENTIONS:
Device: TDCS (Transcranial Direct-current Stimulation) — active TDCS
  Other Names: eldith DC-stimulator (neuroconn, Ilmenau, Germany)
  Arms: Treatment
Device: sham TDCS (Transcranial Direct-current Stimulation) — TDCS at 0mA
  Other Names: eldith DC-stimulator (neuroconn, Ilmenau, Germany)
  Arms: sham

SUMMARY:
The investigators hypothesize that transcranial direct current stimulation over the motor cortex will reduce muscle overflow and improve hand function in children with primary or secondary dystonia.

ELIGIBILITY:
Inclusion Criteria:

* dystonia affecting one or both hands
* age 4 to 21 years

Exclusion Criteria:

* metal implants in the head
* inability to cooperate with instructions

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Hand muscle overflow | 10 minutes post- transcranial Direct-current Stimulation (TDCS)
  surface EMG measure of overflow into muscles during attempted relaxation.

CONTACTS AND LOCATIONS:
Overall Officials: Terence Sanger, MD, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States